CLINICAL TRIAL: NCT06894134
Title: Team-based Learning Intervention in Adolescents to Prevent Risk Factors for Chronic Diseasers - a Cluster Randomized Controlled Trial
Brief Title: Team-based Learning Intervention to Prevent Risk Factors for Chronic Diseases - a Cluster Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, João Guilherme Bezerra Alves, Coordinator, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMIP
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Obesity Prevention; Sedentary Behaviors; Sleep Perception; Alcohol Abuse; Drug Abuse; Physical Inactivity
Keywords: team-based learning; adolescents; prevention; chronic diseases
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior; Alcoholism; Substance-Related Disorders; Chronic Disease

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled trial (cRCT) will be conducted in public schools in Palmares, Brazil, targeting high school students aged 15-19 years. Fourteen schools will be randomly assigned to intervention and control groups. The intervention, consisting of four TBL modules, will cover healthy eating, physical activity, screen time, sleep, tobacco, and alcohol use, delivered by graduate nursing students under faculty supervision. Data collection will take place at three time points: pre-intervention, post-intervention, and three months later. The control group will continue receiving standard health education. Primary outcomes will assess behavioral changes, while secondary outcomes will analyze body mass index (BMI) and blood pressure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adolescent students intervention (Experimental): Students adolescent from Plamares public schools, aging 15 to 19 years who will be submitted to a team-based learning method to provide knowledge to prevent chronic diseases at adult life providing health behaviours.
  Interventions: Other: Team-based learning
- Control (No Intervention): Students adolescent from Palmares aging 15 to 19 years who will receive no education intervention

INTERVENTIONS:
Other: Team-based learning — The intervention will include 4 two-hour modules assessing healthy diet, physical activity and screen time, regular sleep, and tobacco and alcohol use. Each module has specific learning objectives (attachment 1). The TBL is a structured active learning approach that fosters collaboration, critical thinking, and accountability. Each module will involve four key steps: (1) Preparation Phase, where students independently will review pre-class materials to build foundational knowledge; (2) Readiness Assurance Process (RAP), which assesses understanding through an individual quiz (iRAT), a team quiz (tRAT), and an instructor-led clarification session; (3) Application Activities
  Arms: Adolescent students intervention

SUMMARY:
Background: Chronic diseases, such as cardiovascular diseases, diabetes, and cancer, are a major global health issue. Their modifiable risk factors, including poor diet, physical inactivity, irregular sleep, tobacco use, and excessive alcohol consumption, often emerge during adolescence and persist into adulthood. Early educational interventions can promote healthy habits and reduce their prevalence. Team-Based Learning (TBL), an active teaching method, has demonstrated effectiveness in improving knowledge and behaviors essential for a healthy lifestyle. Objective: evaluate whether a TBL-based educational intervention can improve adolescents' knowledge and habits related to chronic disease risk factors. Methods: A cluster randomized controlled trial (cRCT) will be conducted in public schools in Palmares, Brazil, targeting high school students aged 15-19 years. Fourteen schools will be randomly assigned to intervention and control groups. The intervention, consisting of four TBL modules, will cover healthy eating, physical activity, screen time, sleep, tobacco, and alcohol use, delivered by graduate nursing students under faculty supervision. Data collection will take place at three time points: pre-intervention, post-intervention, and three months later. The control group will continue receiving standard health education. Primary outcomes will assess behavioral changes, while secondary outcomes will analyze body mass index (BMI) and blood pressure. Analysis: Data will be analyzed using SPSS, with descriptive statistics, paired and unpaired t-tests, ANOVA, and chi-square tests. The analysis will account for clustering and be conducted using intention-to-treat analysis. Statistical significance will be set at p<0.05. Conclusion: The study will provide evidence on TBL as a scalable tool for preventing risk factors in adolescents, contributing to long-term public health benefits.

DETAILED DESCRIPTION:
Introduction Chronic diseases are leading causes of mortality worldwide, affecting both developed and developing countries. Chronic diseases include cardiovascular diseases, diabetes, stroke, cancer and mental diseases. These diseases have been and continue to be the major causes of worldwide morbidity. They significantly strain healthcare systems and contribute to reduce quality of life and workforce productivity. The estimated cost of chronic disease is expected to reach $47 trillion worldwide by 2030.

Modifiable risk factor for chronic diseases are unhealthy diet, physical inactivity and sedentary behavior, irregular sleep, tobacco use, and excessive alcohol consumption. These risk factors usually begin during childhood and adolescence and persist into adulthood. This age period is critical as they become more exposed to external influences, including peers, media, and their environment, while developing autonomy in decision-making. Intervening during these formative years is essential to promote healthier behaviors and prevent chronic diseases in adulthood.

Some studies on educational interventions for adolescents to prevent chronic disease risk factors have demonstrated promising outcomes in different countries. The Health4Life program, which uses web-based modules to address risk factors, showed increased student engagement and knowledge retention. Another study highlighted the importance of combining education with parental and community involvement to achieve more sustainable behavioral changes. However, other studies including systematic review report limited or no significant changes in healthy behaviors.

Team-based learning (TBL) is an active teaching method with a student-centered approach in which students learn about a subject by working in groups to solve an open-ended problem. This educational approach has several advantages compared to the usual education provided by school teachers, such as improved engagement and active learning andencouragement ofcritical thinking and problem-solving skills.By working in teams, students develop collaboration and communication skills, receive immediate feedback, peer learning, andincrease their motivation, accountability and self-confidence. By presenting real-world problems to solve, TBL also results in better practical knowledge and retention, encourages active engagement and self-directed learning, and fairer assessment of diverse perspectives. TBL appears to be appropriate in improving the knowledge, critical thinking and enhancing their skills and behaviours. The hypothesis that TBL can be use to address risk factors for chronic diseases among adolescents, such as unhealthy diets, physical inactivity, sedentary behavior, irregular sleep patterns, tobacco use, and excessive alcohol consumption, was not tested yet. Studies with education intervention applying the TBL method to adolescents students aiming to preventrisk factor for chronic diseases have not yet been conducted. TBL may contribute to Health Behavior Education enhancingadolescents' understanding of the links between lifestyle choices and health outcomes. TBL may also foster a sense of responsibility and self-efficacy, which are critical for adopting healthier habits. In addition to knowledge, TBL may build skills such as problem-solving, communication, and teamwork, which are vital for sustaining healthy habits into adulthood. Despite its advantages, TBL may present some challenges, such asrequiringmore preparation time for both students and instructors, may be challenging to implement in very large classes, some students may struggle with group dynamics or prefer individual learning styles, and assessment and grading may be more complex compared to traditional methods. However, TBL can offer significant advantages over traditional teaching regarding how we deal with a health problem that potentially affects all adolescent students (a risk factor for chronic diseases), being part of their dailylife, which require practical application of knowledge, collaboration, and the development of real world skills.

Based on all this the objective of this study is to verify if an educational intervention, based on TBL, can prevent risk factors (unhealthy diet, physical inactivity, sedentary behavior, excessive screen time, irregular sleep, tobacco use and excessive alcohol use) for chronic diseases may modify the knowledge and habits of adolescent students.

Methods Study design A cluster randomized controlled trial (cRCT) will be performed using an active learning method, TBL, to prevent risk factors for chronic diseases in adolescent students. A cRCT design reduces the potential for contamination between conditions that would be present were individuals randomized. This project will be previously registered at the ClinicalTrials.gov.

Setting and period The study willl be conducted in the public schools of the city of Palmares, Pernambuco state, Brazil. Palmares has shown a commitment to improving adolescent education through various programs and initiatives. The Basic Education Development Index (IDEB), a key indicator of education quality in Brazil, has increase from 3.9 in 2015 to 4.5 in 2021.Palmares has a population of 54,584 inhabitants (IBGE, 2022), and out of 79 schools, 63 are public and 16 are private. A school year in Brazil runs from March to December with one month vacation (July). The school timings are from 7:30 AM to 11:30 PM in the morning and 1:30 PM to 5:30 PM in the afternoon on working days.

Study participants Data collection After obtaining permission to collect data, the researchers will provide details of the study during the class hour, as well as the inclusion and exclusion criteria to adolescent students. They will also provide information about the study to the school's board. The adolescent students and their parents or legal guardians who agreed to participate in the study will respectively sign an informed assent and an informed consent.

Initially a baseline questionnaire (pre-test) will be applied. This questionnaire (attached) will assess: 1 - Food knowledges, based on the Guidelines for the Brazilian Population (MS), and diet habits; 2 - Benefits of physical activity, based on WHO guidelines, and pattern of physical activity (IPAC); 3 - Knowledge of the association between screen time and health, and determination of participant screen time; 4 - Knowledge of the importance of sleep to the health, and sleep pattern;5 -Knowledge of tobacco and alcohol harms to the health, and identification of habits of cigarette smoking and excessive use of alcohol. We will provide individual students with their own identification number to blind their personal information in the answer sheet both for the clinical reasoning and the socioeconomic status. This same questionnairewill be applied immediately after the end of intervention and three months later.

Randomization The study will randomly select 14 public schools from a list of 63. We will use a computer-generated random number sequence to randomly assign one school to the health-promotion intervention and another to the control intervention within pairs. These randomly selected schools (clusters) will be stratified based on the morning/afternoon turn of the adolescent participants. We will randomly allocate an equal number of clusters from each stratum to the intervention and control arms using stratified random sampling.

Sample size Assuming that the mean and standard deviation of the score in the control group are, respectively, equal to 3 and 1.5 points, it can be seen that two samples, each with 4 classes of 30 students, are sufficient to provide a power of 80% to detect a 50% increase in the mean of the treated group in relation to the control group, assuming a significance level of 5% and an intraclass correlation coefficient of 0.10.

Intervention The goal of the health-promotion intervention is to enhance students' knowledge, attitudes, and skills in maintaining a healthy diet, engaging in physical activity, limiting screen time to less than two hours, maintaining a regular sleep schedule, and abstaining from cigarette smoking and alcohol consumption. This intervention will be based on the active learning method, TBL, a teaching method that uses common real-world problems to promote students' acquisition of knowledge, attitudes, and skills.

Graduate students of a nursing school, under the supervision of their teachers, will apply the intervention. The intervention will include 4 two-hour modules assessing healthy diet, physical activity and screen time, regular sleep, and tobacco and alcohol use. Each module has specific learning objectives (attachment 1). The TBL is a structured active learning approach that fosters collaboration, critical thinking, and accountability. Each module will involve four key steps: (1) Preparation Phase, where students independently will review pre-class materials to build foundational knowledge; (2) Readiness Assurance Process (RAP), which assesses understanding through an individual quiz (iRAT), a team quiz (tRAT), and an instructor-led clarification session; (3) Application Activities, where teams solve real-world problems requiring collaboration, with immediate feedback provided; and (4) Peer Evaluation, ensuring accountability and teamwork improvement. TBL emphasizes permanent teams, problem-based learning, and immediate feedback, promoting deeper comprehension and active engagement.

A healthy diet will be based on the "Dietary Guidelines for the Brazilian Population". Guidelines for physical activity will emanate from WHO. Key recommendations for adolescents include: limit ultra-processed foods, emphasize natural and minimally processed foods, encourage regular meals, including breakfast, hydration, family and social eating practices, food environment awareness. Previous Brazilian studies have shown that many adolescents skip breakfast, have a low consumption of fruits and vegetables, and a high intake of ultra-processed foods. The WHO recommended physical activity guidelines for adolescents; they should engage in at least 60 minutes of moderate-to-vigorous intensity physical activity per day. Regarding screen time we will follow the "Sociedade Brasileira de Pediatria" guidelines: limit screen time to a maximum of 2 to 3 hours per day, always under supervision; they should never "stay up all night" playing games or using electronic devices. The recommendation of the American Academy of Sleep Medicine (AASM)for adolescents to sleep 8 to 10 hours per night regularly will be adopted. Regarding smoking and excessive alcohol consumption the WHO orientations will be followed.

The schools in the control group will provide the usual health education to adolescent students, provided by the municipal education curricula. Teachers of adolescents will complete a questionnaire detailing the scope and structure of any education on risk factors for chronic diseases.

Outcomes The study will primarily measure:(1) the knowledge of healthy dietary habits;(2) the knowledge of the benefits of physical activity and an adoption of a physically active pattern; (3) the knowledge of the health risk of excessive screen time, and the adoption of recreationalscreen time limited to 2 hours per day; (4) the knowledge of health benefits of a regular sleep, and the fulfillment of this habit; (5) the knowledge of the harms of cigarette smoking and excessive alcohol consumption, and abstinence of these unhealthy habits. The knowledge of the adolescent students will be evaluated by a questionnaire based on the bibliography utilized to build the TBL modules and scores, 0 to 10, will be used for each item:health diet, physically active, screen time, sleep regular, smoking and alcohol excess. It will be considered adequate a score equal to or greater than 7.More details are provided in each section on the questionnaire. A healthy dietary habit will be considered adaily consumption of fruits and vegetables, not intake of ultra-processed foods, and not skipping breakfast. The adolescent students will be considered as physically active if they have minimally 150 minutes by week of practicalphysical activity. A sedentary pattern will be considered as a screen time over 2 hours per day. A regular sleep time will be considered as aminimum of 9 hours per day. Regarding smoking and excessive alcohol consumption it will be considered respectively, no smoking and the consumption of more than 60g of pure alcohol per day for men (about 4 standard drinks) and more than 40g for women (about 3 standard drinks).

Secondary outcomes will be behaviors changes in body mass index (kg/m2) and blood pressure (mmHg), among adolescents of both intervention and control arms before, immediately after the intervention and three months later.

Analysis An analysis using the Statistical Package for Social Sciences (SPSS) version 21 will be performed. Intention-to-treat analysis will be used. Descriptive analysis will include the sample mean, standard deviation, and proportions according to the variable types. ANOVA and the chi-square test to compare the statistical significance of continuous and categorical variables will be used. Analyze within-group changes in quantitative variables from baseline to end-line using a paired t-test will be done. Unpaired t-tests to assess between-group comparisons will be applied. In addition to the statistical methods described, a Difference-in-Differences (DID) analysis to control for extraneous changes in both the control and intervention groups over time will be conducted. This analysis will be applied by comparing the pre- and post-intervention differences between groups. The analysis for covariates such as the school shift (morning vs. afternoon) and potential cluster-level variables, including class size and school characteristics, will be adjested. Stratification variables will be incorporated as covariates in the analysis to improve the precision of estimates and account for intra-cluster correlations. A mixed-effects model will be considered to appropriately handle these adjustments. Statistical significance will be set at p<0.05.

Ethical considerations A prior ethical permission from the Ethical Committee on Research at the Instituto de Medicina Integral Prof. Fernando Figueira (IMIP) will be obtained. Permission for the selection of schools by the Secretaria de Educação de Palmares will be also obtained. After informing adolescents and parents about the study purpose, we will achieve their written consent. This is an education intervention study and not involves any potential harm to the study participants.

Declaration of interests The authors have nothing to declare.

Funding sources This work will be supported by the Faculdade de Palmares (FAP), grant number 120300-012025.

Author contributions Conceptualization: JGB Alves; Data curation: JRSJ, YGFFM, CAFLA; Formal analysis: MLU, JGBA; Investigation: JRSJ, YGFFM, CAFLA, ELSS, SBL, SLE; Methodology: JRSJ, YGFFM, MLU, CAFLA, JGBA; Project administration: JRSJ, YGFFM, CAFLA; Supervision: CAFLA; Validation: MLU, SLS; Writing - original draft: JRSJ, MLU, JGBA; Writing - review and editing: JRSJ, YGFFM, MLU, CAFLA, ELSS, SBL, SLS, JGBA.

ATTACHMENT 1 - TEAM-BASED LEARNING (TBL) MODULES FOR HEALTH PROMOTION INTERVENTION

The intervention consists of four structured two-hour modules aimed at addressing key modifiable risk factors for chronic diseases among adolescents. Each module is designed based on Team-Based Learning (TBL) principles, fostering collaboration, problem-solving, and accountability. The modules cover:

1. HEALTHY DIET

   * Learning objectives: Understanding the principles of balanced nutrition, the impact of ultra-processed foods, and the importance of hydration and meal timing.
   * Application: Real-life problem-solving activities related to dietary choices and the consequences of poor nutrition.
2. PHYSICAL ACTIVITY AND SCREEN TIME

   * Learning objectives: Recognizing the benefits of physical activity, understanding WHO recommendations, and evaluating the risks of excessive screen time.
   * Application: Team-based scenarios assessing daily habits, identifying barriers to physical activity, and proposing behavior changes.
3. REGULAR SLEEP PATTERNS

   * Learning objectives: Understanding the role of sleep in overall health, the impact of sleep deprivation, and strategies to improve sleep hygiene.
   * Application: Students analyze their sleep patterns and propose realistic improvements based on scientific evidence.
4. TOBACCO AND ALCOHOL USE

   * Learning objectives: Identifying the health risks of tobacco and excessive alcohol consumption, understanding peer pressure influences, and strategies for prevention.
   * Application: Case studies and team discussions on real-world scenarios involving tobacco and alcohol exposure.

TBL IMPLEMENTATION FRAMEWORK

Each module follows a four-step TBL process:

1. PREPARATION PHASE

   * Students independently review pre-class materials (scientific articles, infographics, videos).
   * Materials align with health education guidelines, ensuring foundational knowledge before class discussions.
2. READINESS ASSURANCE PROCESS (RAP)

   * Students complete Individual Readiness Assurance Tests (iRAT) to assess comprehension.
   * Teams then collaborate on Team Readiness Assurance Tests (tRAT), discussing and defending their answers.
   * An instructor-led review session clarifies misconceptions and reinforces key concepts.
3. APPLICATION ACTIVITIES

   * Teams engage in real-world problem-solving tasks related to the module topic.
   * Activities are designed to encourage critical thinking, peer discussion, and decision-making.
   * Immediate feedback from facilitators ensures concept reinforcement.
4. PEER EVALUATION

   * Students assess their peers' contributions, promoting accountability and teamwork.
   * Feedback mechanisms encourage self-reflection and continuous improvement in collaborative learning.

EDUCATIONAL RATIONALE

TBL is an evidence-based pedagogical approach that enhances student engagement, deepens conceptual understanding, and promotes active learning. By integrating case-based discussions, structured teamwork, and real-world application, the intervention aims to foster long-term behavior changes that reduce the prevalence of chronic disease risk factors in adolescents.

The intervention will be implemented by graduate nursing students under faculty supervision, ensuring methodological consistency and alignment with public health education standards.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent students of high school
* Age ranging from 15 to 19 years old.

Exclusion Criteria:

* Cognitive limitations
* Physical limitations
* Communication limitations
* Use of medications that interfere with eating, physical activity, or sleeping habits.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge and behaviour of healthy dietary habits, physical activity pattern, regular sleep and no tobaco and excessive alcohol | 6 months
  The knowledge of the adolescent students will be evaluated by scores, 0 to 10, for each item:health diet, physically active, screen time, sleep regular, smoking and alcohol excess. It will be considered adequate a score equal to or greater than 7.More details are provided in each section on the questionnaire. A healthy dietary habit will be considered adaily consumption of fruits and vegetables, not intake of ultra-processed foods, and not skipping breakfast. The adolescent students will be considered as physically active if they have minimally 150 minutes by week of practicalphysical activity. A sedentary pattern will be considered as a screen time over 2 hours per day. A regular sleep time will be considered as aminimum of 9 hours per day. Regarding smoking and excessive alcohol consumption it will be considered respectively, no smoking and the consumption of more than 60g of pure alcohol per day for men (about 4 standard drinks) and more than 40g for women (about 3 standard drinks)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.imip.org.br